CLINICAL TRIAL: NCT03478748
Title: The Impact of Anticipatory Guidance on Early Childhood Caries: a Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Norintan Ab Murat, Associate Professor, University of Malaya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DFCO1505/0005P
Record Dates: First submitted 2018-02-26; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Oral health literacy
MeSH Terms: conditions — Dental Caries | interventions — Health Education, Dental

STUDY DESIGN:
Intervention Model Description: The model is an oral health education package that covers the following aspects: (i) cognitive component (for example, the provision of basic oral health knowledge using an anticipatory guidance technique); (ii) psychomotor component (for example, the demonstration of basic oral health skills such as toothbrushing skills with a hands-on practical); and (iii) attitude component (activities that help to improve the children's attitude towards oral health). Children (along with their older siblings and mothers) in the study group were required to make six-monthly visits to the dental clinic in the three-year study period. Those in the control group received the conventional Ministry of Health programme.
Masking Description: Both investigators and participants knew about the intervention and who were involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-to-one dental health education (Active Comparator): Conventional oral health education programme that mainly focuses at child level, which has been the normal practice at the Ministry of Health, were provided to the control participants.
  Interventions: Other: Dental health education
- anticipatory guidance technique (Experimental): Anticipatory guidance technique were applied where appropriate dental health education (according to the children's milestones) were provided to mothers and their children.
  Interventions: Other: Dental health education

INTERVENTIONS:
Other: Dental health education — Anticipatory guidance given to mothers to promote their children's oral health.
  Other Names: Anticipatory guidance

SUMMARY:
This study aimed to compare the impact of anticipatory guidance on the caries incidence of 2-3-year-old preschool children and their 4-6-year-old siblings, as well as on their mothers' oral health literacy, as compared to the conventional Ministry of Health (MOH) programme.

DETAILED DESCRIPTION:
This quasi-experimental study was conducted at two government dental clinics in Batu Pahat District, Malaysia. The samples comprised of 478 mother-child-sibling trios (233 families in the intervention group, and 245 families in the control group). An oral health package named the Family Dental Wellness Programme (FDWP) was designed to provide anticipatory guidance to the intervention group at six-month intervals over three years. The control group received the standard MOH oral health education activities. The impact of FDWP on net caries increment, caries prevented fraction, and mother's oral health literacy was assessed after three years of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 2-3 years old
* Older sibling aged 4 to 6 years categorized as having high caries risk based on a Caries Risk Assessment tool adapted from the American Association of Paediatric Dentistry
* Mothers who were willing to participate in the study

Exclusion Criteria:

• Medically compromised children

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 478 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of dental caries | Baseline and 3 years
  Change from baseline dental caries prevalence at 3 years using visual and tactile examination

SECONDARY OUTCOMES:
Mothers' oral health literacy | Baseline and 3 years
  Changes in mothers' oral health literacy at 3 year follow up using a validated Dental Health Literacy instruments

CONTACTS AND LOCATIONS:
Overall Officials: Norintan Ab Murat, PhD, Study Chair — University of Malaya
Locations (1):
- Batu Pahat Dental Clinic, Batu Pahat, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ismail A, Razak IA, Ab-Murat N. The impact of anticipatory guidance on early childhood caries: a quasi-experimental study. BMC Oral Health. 2018 Jul 27;18(1):126. doi: 10.1186/s12903-018-0589-0. PMID 30053849